CLINICAL TRIAL: NCT04913051
Title: Interest of Day Hospital Care for Patients With Chronic Regional Pain Syndrome Referred to the Chronic Pain Unit for the First Time
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier le Mans (Other)
Responsible Party: Sponsor
Other Study IDs: CHM-2020/S44/15
Record Dates: First submitted 2021-05-21; First posted 2021-06-04 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-05

CONDITIONS: Chronic Regional Pain Syndrome
Keywords: Chronic Regional Pain Syndrome; day hospital; Chronic Pain Unit
MeSH Terms: conditions — Complex Regional Pain Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Chronic Regional Pain Syndrome (CRPS) is a chronic disabling disease. Patients present a variable picture associating pain localized to an articular or peri-articular region, motor and vasomotor disorders and trophic disorders.

Its pathophysiology, still poorly understood to this day, results from local inflammatory phenomena complicated by peripheral sensitization and central spinal and cerebral sensitization.

The diagnosis is made difficult by the fluctuating nature of the symptoms and the absence of specific complementary examination.

The treatment of CRPS is symptomatic and requires multidisciplinary care. CRPS is responsible for an alteration in the patient's quality of life. This pathology has a global impact because it affects not only the biomedical sphere but also the socio-family, professional and psychological spheres.

The investigators hypothesize that multidisciplinary intervention in the Day Hospital would improve the quality of life of patients with CRPS. The investigators also think that the passage in Day Hospital would make it possible to improve the pains, the functionality of the affected limb as well as the satisfaction of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient volunteers over 18 years of age
* Diagnosis of CRPS according to the Budapest criteria
* Referred to pain assessment and treatment center

Exclusion Criteria:

* Patients unable to express their wishes or understand the protocol
* Diagnosis of CRPS not meeting Budapest criteria
* Patients previously seen at pain assessment and treatment center for the care of CRPS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Chronic Regional Pain Syndrome referred to the Chronic Pain Facility for the first time
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-05-20 (Actual); Primary Completion 2023-05-20 (Estimated); Study Completion 2023-05-20 (Estimated)

PRIMARY OUTCOMES:
Evaluate impact of day hospital care on quality of life | 3 months after day hospital
  Impact of quality of life was assessed by questionnaire Short Form Health Survey (SF36). A score ranging from 0 to 100 is obtained. A low score reflects a perception of poor health, loss of function, presence of pain.
Evaluate impact of day hospital care on quality of life | 6 months after day hospital
  Impact of quality of life was assessed by questionnaire Short Form Health Survey (SF36). A score ranging from 0 to 100 is obtained. A low score reflects a perception of poor health, loss of function, presence of pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Du Mans, Le Mans, France

IPD SHARING:
Plan to Share IPD: No